CLINICAL TRIAL: NCT03103451
Title: A Comparative Randomized Single-Blind Placebo-controlled Study of the Pharmacokinetics, Pharmacodynamics, Tolerability, and Safety of Single Escalating Subcutaneous Doses of BCD 121 in Healthy Volunteers
Brief Title: First-in-human Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Various Doses of BCD-121 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BCD-121-1
Record Dates: First submitted 2017-03-27; First posted 2017-04-06 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): This cohort includes 3 subjects in BCD-121 group and 1 subject in placebo group.
  Intervention: BCD-121/ placebo
  Interventions: Drug: BCD-121; Other: Placebo
- Cohort 2 (Experimental): This cohort includes up to 6 subjects in BCD-121 group and 1 subject in placebo group.
  Intervention: BCD-121/ placebo
  Interventions: Drug: BCD-121; Other: Placebo
- Cohort 3 (Experimental): This cohort includes up to 6 subjects in BCD-121 group and 1 subject in placebo group.
  Intervention: BCD-121/ placebo
  Interventions: Drug: BCD-121; Other: Placebo
- Cohort 4 (Experimental): This cohort includes up to 6 subjects in BCD-121 group and 1 subject in placebo group.
  Intervention: BCD-121/ placebo
  Interventions: Drug: BCD-121; Other: Placebo
- Cohort 5 (Experimental): This cohort includes up to 6 subjects in BCD-121 group and 1 subject in placebo group.
  Intervention: BCD-121/ placebo
  Interventions: Drug: BCD-121; Other: Placebo
- Cohort 6 (Experimental): This cohort includes up to 6 subjects in BCD-121 group and 1 subject in placebo group.
  Intervention: BCD-121/ placebo
  Interventions: Drug: BCD-121; Other: Placebo
- Cohort 7 (Experimental): This cohort includes up to 6 subjects in BCD-121 group and 1 subject in placebo group.
  Intervention: BCD-121/ placebo
  Interventions: Drug: BCD-121; Other: Placebo

INTERVENTIONS:
Drug: BCD-121
  Other Names: monoclonal bispecific antibody against human IL-17/ TNFa
Other: Placebo

SUMMARY:
This is an open label, phase 1, "3+3", placebo-controlled dose escalating study of tolerability, safety, pharmacokinetics, pharmacodynamics and immunogenicity of a single subcutaneous injection of the novel monoclonal bispecific antibody against human IL-17/TNFa. The study will enroll 28 healthy male volunteers.

DETAILED DESCRIPTION:
Simultaneous blockade of IL-17 and TNFa is a potential therapeutic way of treatment of several autoimmune disorders. BCD-121 is a novel humanized monoclonal bispecific antibody against human IL17 and TNFa developed by JCS BIOCAD (Russia) which is now on the first step of clinical evaluation. BCD-121-1 study is the first-in-human clinical trial which is intended to evaluate tolerability, safety, pharmacokinetics, pharmacodynamics and immunogenicity of BCD-121 when used as a single step-by-step escalating subcutaneous dose in healthy male volunteers. During this study it is expected to determine diapason of safety doses of BCD-121 (incl. MTD) which thereafter can be evaluated in phase 2 studies.

ELIGIBILITY:
Inclusion Criteria:

* singed informed consent
* male gender
* 18-45 years of age inclusively
* BMI between18.5-30.0 kg/sq.m.
* absence of any sings of hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality at screening or/and in anamnesis
* parameters of complete blood count, blood biochemistry, and urinalysis do not exceed reference values, which are used at Study site laboratory
* normal hemodynamic parameters
* absence of chronic infections (HIV, syphilis, hepatitis В or С, tuberculosis ) and chronic inflammation
* absence of infections within 4 weeks before randomization
* absence of mental disorders or other conditions (incl. depression), which may affect the ability of participant to follow Protocol
* health well-being (by volunteer's opining opinion) for at least 30 days before randomization.
* absence of alcohol or drug addiction signs (incl. history of such addiction)
* volunteer's ability to follow Protocol procedures
* consent of volunteers and their sexual partners with childbearing potential to use adequate contraception

Exclusion Criteria:

* history of use of monoclonal antibodies against IL-17 or TNFa
* known severe allergy (anaphylaxis or multidrug intolerance)
* known intolerance to medicines containing monoclonal antibodies (murine, humanized, human) or to any excipients of BCD-121/placebo
* major surgery within 30 days prior screening
* severe infections (required hospitalization, parenteral use of antimicrobial agents)
* systemic use of antimicrobials
* more than 4 episodes of respiratory tract infections within 6 months prior the screening
* presence of any disorders which may affect pharmacokinetics of BCD-121
* history of fever which was equal or exceeded 40 degrees in Celsius
* history of hepatic transaminases increase 2.5 x ULN
* history of seizures
* actual or prior depression, suicidal tendencies
* use of any medicines, vitamins, biologically active additives within 14 days prior the date of BCD-085 injection
* use of any medicines which affects hemodynamics or hepatic function within 30 days prior the date of BCD-121 injection
* simultaneous participation in any other clinical trial, as well as former participation in other clinical trials within 3 months before this study initiation.
* previous participation in this study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration of BCD-121-time Curve From Zero (0) Hours to 2160 Hours After the Single Subcutaneous Injection of BCD-121 | 90 days

SECONDARY OUTCOMES:
Maximum Concentration of BCD-121 After Single Subcutaneous Injection | 90 days
Time to Maximum Concentration of BCD-121 After Single Subcutaneous Injection | 90 days